CLINICAL TRIAL: NCT04445623
Title: Prasugrel in the Prevention of Severe SARS-CoV2 Pneumonia in Hospitalised Patients
Brief Title: Prasugrel in Severe COVID-19 Pneumonia
Acronym: PARTISAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MGI-COVID-19-prasugrel
Record Dates: First submitted 2020-06-04; First posted 2020-06-24 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-05

CONDITIONS: COVID19; Thrombosis
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — Prasugrel Hydrochloride; Tablets

STUDY DESIGN:
Intervention Model Description: Experimental phase 3 drug trial, randomized 1:1, double-blind, multicentre in patients treated with prasugrel vs placebo.
Who Masked: Participant, Care Provider
Masking Description: use of placebo tablets of the same shape, colour of the investigational drug. Identical time and route of administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prasugrel hydrochloride (Active Comparator): film-coated tablets of prasugrel hydrochloride (10 mg daily dose after loading dose of 60 mg)
  Interventions: Drug: Prasugrel Hydrochloride 10 MG Oral Tablet
- placebo (Placebo Comparator): film-coated tablets of placebo (10 mg daily dose after loading dose of 60 mg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasugrel Hydrochloride 10 MG Oral Tablet — administration of prasugrel daily for 15 days
  Arms: prasugrel hydrochloride
Drug: Placebo — administration of placebo daily for 15 days
  Arms: placebo

SUMMARY:
Inflammatory diseases favour the onset of venous thromboembolic events in hospitalized patients. Thromboprophylaxis with a fixed dose of heparin/low molecular weight heparin (LMWH) is recommended if concomitant inflammatory disease. In severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) pneumonia an inflammation-dependent thrombotic process occurs and platelet activation may promote thrombosis and amplify inflammation, as indicated by previous experimental evidence , and the similarities with atherothrombosis and thrombotic microangiopathies. Antiplatelet agents represent the cornerstone in the prevention and treatment of atherosclerotic arterial thromboembolism, with limited efficacy in the context of venous thromboembolism. The use of purinergic receptor P2Y12 inhibitors in pneumococcal pneumonia may improve inflammation and respiratory function in humans. There are no validated protocols for thrombosis prevention in Covid-19. There is scientific rationale to consider a P2Y12 inhibitor for the prevention of thrombosis in the pulmonary circulation and attenuation of inflammation. This is supported by numerous demonstrations of the anti-inflammatory activity of P2Y12 inhibitors and the evidence of improvement in respiratory function both in human and experimental pathology. Prasugrel could be considered as an ideal candidate drug for Covid-19 patients because of higher efficacy and limited Interactions with drugs used in the treatment of Sars-CoV2. The hypothesis underlying the present study project is that in Covid-19 platelet activation occurs through an inflammation-dependent mechanism and that early antithrombotic prophylaxis in non-critical patients could reduce the incidence of pulmonary thrombosis and respiratory and multi-organ failure improving clinical outcome in patients with SARS-CoV2 pneumonia. The prevention of thrombogenic platelet activity with a P2Y12 inhibitor could be superior to fixed dose enoxaparin alone. The proposed treatment is feasible in all coronavirus disease 2019 (COVID-19) patients, regardless of the treatment regimen (antivirals, anti-inflammatory drugs, antibiotics), except for specific contraindications.

DETAILED DESCRIPTION:
Severe respiratory failure and multi-organ damage in coronavirus disease 2019 (COVID-19) patients have not a unitary pathophysiological interpretation. There is evidence of an association between the clinical entity of the disease and its severity with the plasma levels of D-dimer and inflammatory indexes. On the basis of retrospective investigations there is accumulating evidence of alterations in the haemostatic parameters that with increased D-dimer values, increased coagulation time and platelets may be predictors of worse prognosis. A systematic survey conducted in the coronavirus disease 2019 (COVID-19) Centre of the AOUI Verona, as part of the Database and Study on the role of platelets in the clinical manifestations of COVID-19 (Ethics Committee CESC Verona and Rovigo approved) revealed by means of computerized tomography (CT) angiograph in patients with a persistent respiratory deficit and very high D-dimer values mainly multiple, bilateral vascular occlusions involving the segmental and subsegmental branches of the pulmonary arteries. This finding is suggestive of a frequent and clinically relevant thrombotic process in a appreciable number (approximately 20%) of patients with COVID-19 pneumonia hospitalized in medical wards. It is a well-established clinical notion that acute and chronic inflammatory diseases may favour the onset of venous thromboembolic events in hospitalized patients. Thromboprophylaxis with a fixed dose of heparin/low molecular weight heparin (LMWH) is recommended for medical patient with concomitant neoplasia or inflammatory disease. It is conceivable that under conditions, such as SARS-CoV2 pneumonia, an inflammation-dependent thrombotic process takes place and that platelet activation may play a pathogenic role both in the thrombotic process and in the amplification of the inflammatory process. In fact, there is experimental evidence that platelet activation in inflammation would lead to accelerated coagulation and a thrombotic vascular occlusion, with similarities to what is widely documented in atherothrombosis and thrombotic microangiopathies. The administration of antiplatelet drugs represents the cornerstone for the prevention and treatment of arterial thromboembolism in atherosclerotic disease and has also shown some limited efficacy also in the context of venous and arterial thromboembolism associated with atrial fibrillation. Preliminary observations indicate that the use of purinergic receptor P2Y12 inhibitors during pneumococcal pneumonia may improve the inflammatory process and respiratory function in humans. There are currently no validated protocols for thrombosis prevention in the field of pulmonary viral diseases, in particular COVID-19. There is adequate scientific rationale to consider the use of a P2Y12 inhibitor antiplatelet drug for the prevention of thrombosis in the pulmonary circulation and the attenuation of pulmonary inflammation. The use of a P2Y12 inhibitor is motivated by numerous experimental demonstrations of the anti-inflammatory activity of P2Y12 inhibitors and by the evidence of improvement of respiratory function parameters both in humans and experimental models. Prasugrel could be considered as an ideal candidate drug for administration in Covid-19 patients because of its higher efficacy in acute coronary syndrome compared to clopidogrel. Interactions of prasugrel with drugs used for the treatment of SARS-CoV2 are limited. The hypothesis underlying the present study project is that in Covid-19 platelet activation occurs via an inflammation-dependent mechanism and that early antithrombotic prophylaxis in non-critical patients, like those admitted to medical wards, could reduce the incidence of pulmonary thrombosis as well as respiratory and multi-organ failure, contributing to improve clinical outcome of the patients with pneumonia caused by SARS-CoV2 viruses. The anticoagulant activity exerted by a fixed dose of enoxaparin (4000U/day), recommended in patients with the clinical features described, according to a note of the "Italian Medicines Agency" (AIFA), together with the prevention of thrombogenic activity of platelets by means of a P2Y12 inhibitor could prevent aggravation of COVID-19 patients to a greater extent than enoxaparin alone given at the same dose. Early initiation of treatment should mitigate the presentation of pneumonia. The proposed treatment is feasible in all COVID-19 patients, regardless of the treatment regimen used for their condition (antivirals, anti-inflammatory drugs, antibiotics), except for specific contraindications to the use of prasugrel, or placebo if patients are treated with antiplatelet drugs.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 pneumonia
* Age over 18 years
* Willingness to express consent

Exclusion Criteria:

* Active neoplasia or in maintenance therapy
* Pregnancy and breastfeeding
* Any absolute contraindication to the use of antiplatelet drugs
* Pathological bleeding in progress.
* Recent major bleeding at any location
* Need to use therapeutic doses of oral anticoagulants or heparins
* Need to use antiplatelet in combination for clinical indication
* Hypersensitivity to the active substance prasugrel or any of the excipients
* Clinical history of stroke or transient ischemic attack (TIA).
* Severe liver failure (Child-Pugh class C).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
P/F ratio at day 7 | day 7
  PaO2/FiO2 ratio (arterial oxygen tension divided by the fraction of inspired oxygen) detected after 7 days of treatment

SECONDARY OUTCOMES:
Daily P/F ratio | 15 days
  PaO2/FiO2 ratio (arterial oxygen tension divided by the fraction of inspired oxygen) detected daily for 15 days
Daily need for oxygen supply | 15 days
  daily need for oxygen supply for 15 days
Need for ICU | day 15 and day 30
  Number of patients requiring transfer to the intensive care unit (ICU) by treatment arm
Death | 15 day and day 30
  death by day 15 and day 30 by treatment arm
MOF | day 15 and day 30
  Multi-organ failure (MOF) by day 15 and day 30 assessed using sequential organ failure assessment score (SOFA) score (Units 0-4 better outcome, over 30 worse outcome) by treatment arm
Discharge | day 15 and day 30
  Number of patients discharged after improvement by day 15 and day 30 by treatment arm
Clinical progression of the disease SOFA score | day 15 and day 30
  Clinical progression of the disease evaluated by SOFA score (Units 0-6 better outcome, 15-24 worse outcome) by day 15 and day 30
Clinical progression of the disease APACHE II | day 15 and day 30
  Clinical progression of the disease evaluated by Acute Physiology And Chronic Health Evaluation (APACHE II) score (Units 1-5 better outcome, over 30 worse outcome) by day 15 and day 30
Venous thrombosis/ pulmonary embolism/thrombosis | day 15 and day 30
  Number of patients with venous thrombosis/ pulmonary embolism/thrombosis by day 15 and day 30
Need for CT imaging | day 15
  Number of patients requiring computerized tomography (CT) imaging due to worsening of respiratory function by treatment arm
Daily Temperature | 15 days
  Body temperature measured twice daily for 15 days, C°
Daily blood pressure | 15 days
  Blood pressure measured twice daily for 15 days, mmHg
Daily total blood count Hemoglobin | 15 days
  Total blood count measured in venous blood for 15 days, Hemoglobin, g/L (cell/mcL
Daily total blood count Red Blood Cells | 15 days
  Total blood count measured in venous blood for 15 days, Red Blood cells (cell/mcL)
Daily total blood count Leukocytes | 15 days
  Total blood count measured in venous blood for 15 days, Leukocytes (cell/mcL)
Daily total blood count Platelets | 15 days
  Total blood count measured in venous blood for 15 days, platelets (cell/mcL)
Daily indices of organ damage Liver | 15 days
  ALT U/L in venous blood
Indices of inflammation C-reactive protein | day 1, 2, 7, 15
  C-reactive protein microg/L in venous blood
Indices of haemostasis PT | day 1, 2, 7,15
  PT ratio in venous blood by treatment arm
Daily progression at imaging (chest-X-ray) | 15 days
  progression of lung infiltrates as detected by chest-X-ray by treatment arm
Major bleeding | day 1, 2, 7, 15, 30
  Major and/or clinically relevant bleeding according to International Society of Thrombosis and Haemostasis (ISTH) bleeding scale (Unit 0 better outcome, 4 worse outcome, 11 items) during treatment.
Total bleeding | day 1, 2, 7, 15, 30
  Total bleeding according to International Society of Thrombosis and Haemostasis (ISTH bleeding) scale (Unit 0 better outcome, 4 worse outcome, 11 items) during treatment.
Unexpected clinical or laboratory findings | day 1, 2, 7, 15
  Number of unexpected changes in clinical or laboratory findings not included in the predefined list of outcomes during treatment. .
Indices of inflammation D-dimer | day 1, 2, 7, 15
  D-dimer microg/L in venous blood
Indices of inflammation Fibrinogen | day 1, 2, 7, 15
  Fibrinogen g/L in venous blood
Indices of inflammation IL-6 | day 1, 2, 7, 15
  Interleukin (IL)-6 pg/mL in venous blood by treatment arm
Indices of inflammation IL-1 | day 1, 2, 7, 15
  Interleukin (IL)-1 pg/mL in venous blood by treatment arm
Daily indices of organ damage kidney | 15 days
  serum creatinine micromol/L by treatment arm
Daily indices of organ damage heart | 15 days
  troponin t ng/L by treatment arm
Haemostasis aPTT | day 1, 2, 7,15
  aPTT ratio by treatment arm
Haemostasis VASP PRI | day 1, 2, 7,15
  Vasodilator stimulated phosphoprotein (VASP) phosphorylation (PRI) % by treatment arm
Haemostasis platelet-leukocytes aggregates | day 1, 2, 7,15
  Platelet-leukocytes aggregates % in peripheral by treatment arm

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

REFERENCES:
- [Background] Obi AT, Tignanelli CJ, Jacobs BN, Arya S, Park PK, Wakefield TW, Henke PK, Napolitano LM. Empirical systemic anticoagulation is associated with decreased venous thromboembolism in critically ill influenza A H1N1 acute respiratory distress syndrome patients. J Vasc Surg Venous Lymphat Disord. 2019 May;7(3):317-324. doi: 10.1016/j.jvsv.2018.08.010. Epub 2018 Nov 23. PMID 30477976
- [Background] Smeeth L, Cook C, Thomas S, Hall AJ, Hubbard R, Vallance P. Risk of deep vein thrombosis and pulmonary embolism after acute infection in a community setting. Lancet. 2006 Apr 1;367(9516):1075-1079. doi: 10.1016/S0140-6736(06)68474-2. PMID 16581406
- [Background] Margraf A, Zarbock A. Platelets in Inflammation and Resolution. J Immunol. 2019 Nov 1;203(9):2357-2367. doi: 10.4049/jimmunol.1900899. PMID 31636134
- [Background] Eck RJ, Bult W, Wetterslev J, Gans ROB, Meijer K, van der Horst ICC, Keus F. Low Dose Low-Molecular-Weight Heparin for Thrombosis Prophylaxis: Systematic Review with Meta-Analysis and Trial Sequential Analysis. J Clin Med. 2019 Nov 21;8(12):2039. doi: 10.3390/jcm8122039. PMID 31766453
- [Background] Jackson SP, Darbousset R, Schoenwaelder SM. Thromboinflammation: challenges of therapeutically targeting coagulation and other host defense mechanisms. Blood. 2019 Feb 28;133(9):906-918. doi: 10.1182/blood-2018-11-882993. Epub 2019 Jan 14. PMID 30642917
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Becattini C, Agnelli G, Schenone A, Eichinger S, Bucherini E, Silingardi M, Bianchi M, Moia M, Ageno W, Vandelli MR, Grandone E, Prandoni P; WARFASA Investigators. Aspirin for preventing the recurrence of venous thromboembolism. N Engl J Med. 2012 May 24;366(21):1959-67. doi: 10.1056/NEJMoa1114238. PMID 22621626
- [Background] Simes J, Becattini C, Agnelli G, Eikelboom JW, Kirby AC, Mister R, Prandoni P, Brighton TA; INSPIRE Study Investigators (International Collaboration of Aspirin Trials for Recurrent Venous Thromboembolism). Aspirin for the prevention of recurrent venous thromboembolism: the INSPIRE collaboration. Circulation. 2014 Sep 23;130(13):1062-71. doi: 10.1161/CIRCULATIONAHA.114.008828. Epub 2014 Aug 25. PMID 25156992
- [Background] Sexton TR, Zhang G, Macaulay TE, Callahan LA, Charnigo R, Vsevolozhskaya OA, Li Z, Smyth S. Ticagrelor Reduces Thromboinflammatory Markers in Patients With Pneumonia. JACC Basic Transl Sci. 2018 Aug 28;3(4):435-449. doi: 10.1016/j.jacbts.2018.05.005. eCollection 2018 Aug. PMID 30175268
- [Background] Rudolph TK, Fuchs A, Klinke A, Schlichting A, Friedrichs K, Hellmich M, Mollenhauer M, Schwedhelm E, Baldus S, Rudolph V. Prasugrel as opposed to clopidogrel improves endothelial nitric oxide bioavailability and reduces platelet-leukocyte interaction in patients with unstable angina pectoris: A randomized controlled trial. Int J Cardiol. 2017 Dec 1;248:7-13. doi: 10.1016/j.ijcard.2017.06.099. Epub 2017 Jul 1. PMID 28709700
- [Background] Johnston LR, La Flamme AC, Larsen PD, Harding SA. Prasugrel inhibits platelet-enhanced pro-inflammatory CD4+ T cell responses in humans. Atherosclerosis. 2015 Mar;239(1):283-6. doi: 10.1016/j.atherosclerosis.2015.01.006. Epub 2015 Jan 14. PMID 25635327
- [Background] Totani L, Dell'Elba G, Martelli N, Di Santo A, Piccoli A, Amore C, Evangelista V. Prasugrel inhibits platelet-leukocyte interaction and reduces inflammatory markers in a model of endotoxic shock in the mouse. Thromb Haemost. 2012 Jun;107(6):1130-40. doi: 10.1160/TH11-12-0867. Epub 2012 Mar 22. PMID 22436970
- [Background] Ancrenaz V, Deglon J, Samer C, Staub C, Dayer P, Daali Y, Desmeules J. Pharmacokinetic interaction between prasugrel and ritonavir in healthy volunteers. Basic Clin Pharmacol Toxicol. 2013 Feb;112(2):132-7. doi: 10.1111/j.1742-7843.2012.00932.x. Epub 2012 Oct 5. PMID 22900583
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Yin S, Huang M, Li D, Tang N. Difference of coagulation features between severe pneumonia induced by SARS-CoV2 and non-SARS-CoV2. J Thromb Thrombolysis. 2021 May;51(4):1107-1110. doi: 10.1007/s11239-020-02105-8. PMID 32246317
- [Background] Minuz P, Mansueto G, Mazzaferri F, Fava C, Dalbeni A, Ambrosetti MC, Sibani M, Tacconelli E. High rate of pulmonary thromboembolism in patients with SARS-CoV-2 pneumonia. Clin Microbiol Infect. 2020 Nov;26(11):1572-1573. doi: 10.1016/j.cmi.2020.06.011. Epub 2020 Jun 18. No abstract available. PMID 32565320
- [Background] Cattaneo M, Bertinato EM, Birocchi S, Brizio C, Malavolta D, Manzoni M, Muscarella G, Orlandi M. Pulmonary Embolism or Pulmonary Thrombosis in COVID-19? Is the Recommendation to Use High-Dose Heparin for Thromboprophylaxis Justified? Thromb Haemost. 2020 Aug;120(8):1230-1232. doi: 10.1055/s-0040-1712097. Epub 2020 Apr 29. No abstract available. PMID 32349132
- [Background] Sjalander A, Jansson JH, Bergqvist D, Eriksson H, Carlberg B, Svensson P. Efficacy and safety of anticoagulant prophylaxis to prevent venous thromboembolism in acutely ill medical inpatients: a meta-analysis. J Intern Med. 2008 Jan;263(1):52-60. doi: 10.1111/j.1365-2796.2007.01878.x. PMID 18088252
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818